CLINICAL TRIAL: NCT06399900
Title: ENhancing Exercise with LIGHT to Improve Functioning in PAD: the ENLIGHTEN PAD Trial
Brief Title: ENhancing Exercise with LIGHT to Improve Functioning in PAD
Acronym: ENLIGHTEN PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00219103
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Aging; Walking, Difficulty
Keywords: light therapy; peripheral artery disease; exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Thirty-two participants with PAD will be randomized to either 660 nm light + home-based exercise or sham light + home-based exercise for four months. Both groups will receive the same home-based high intensity walking exercise intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This will be a double blinded study where both the participant and the people collecting data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Far red light therapy + home-based walking exercise (Experimental): Subgroup of participants receiving home-based walking exercise and the 670 nm far red light device
  Interventions: Device: Far red light therapy; Behavioral: Home-based walking exercise
- Sham therapy + home-based walking exercise (Sham Comparator): Subgroup of participants receiving home-based walking exercise and the sham light device, far red light device covered with blue filter paper to block 670 nm light, resulting in mean power generated of 0.24 mW/cm2, compared to 26.3 mW/cm2 for the intervention, a 100-fold difference.
  Interventions: Device: Sham light therapy; Behavioral: Home-based walking exercise

INTERVENTIONS:
Device: Far red light therapy — All participants will receive one far red light device per leg. Participants will be asked to use their two light devices daily, exposing their bare legs to the devices for 10 minutes twice per day. An unblinded study coordinator will deliver the light devices to each participant's home, positioning the devices 15 cm behind the participant's heels, using tape on the floor to mark where the light and feet should be positioned. Twice each day, the participant flips a switch on the device to begin each session. A timer will turn off the device after 10 minutes. A power meter will measure the total time that the device was turned on. Participants will also record use of the light in a log.
  Arms: Far red light therapy + home-based walking exercise
Device: Sham light therapy — All participants will receive one sham device per leg. Participants will be asked to use their two light devices daily, exposing their bare legs to the devices for 10 minutes twice per day. An unblinded study coordinator will deliver the light devices to each participant's home, positioning the devices 15 cm behind the participant's heels, using tape on the floor to mark where the light and feet should be positioned. Twice each day, the participant flips a switch on the device to begin each session. A timer will turn off the device after 10 minutes. A power meter will measure the total time that the device was turned on. Participants will also record use of the light in a log.
  Arms: Sham therapy + home-based walking exercise
Behavioral: Home-based walking exercise — This study involves a 16 week intervention where participants will walk at home for exercise with guidance from a study coach. Participants will have 4 in-person visits in the first four weeks and then have weekly phone calls in the last 12 weeks of the intervention with their coach.

SUMMARY:
The ENLIGHTEN PAD Trial will collect preliminary data to test whether daily 660 nm light treatment of the lower extremities immediately before home-based walking exercise sessions improves six-minute walk distance at 4-month follow-up, compared to sham light, in people with lower extremity peripheral artery disease (PAD).

DETAILED DESCRIPTION:
The ENLIGHTEN PAD Trial will collect preliminary data to test whether daily 660 nm light treatment of the lower extremities immediately before home-based walking exercise sessions improves six-minute walk distance at 4-month follow-up, compared to sham light, in people with lower extremity peripheral artery disease (PAD) (Primary Aim #1). In Primary Aim #2, the investigators will measure the acute effect of the first treatment of 660 nm light on six-minute walk distance and on walking intensity (measured with the ActiGraph accelerometer) during the six-minute walk. In secondary and exploratory aims, the investigators will delineate biologic pathways by which 660 nm light enhances the benefits of home-based walking exercise, by measuring the effects of 660 nm light on exercise intensity during the exercise intervention and by measuring the effects of 660 nm light on plasma nitrosothiols, leg perfusion, and gastrocnemius muscle health and mitochondrial activity. Exercise intensity will be measured by the well validated ActiGraph accelerometer.

The ENLIGHTEN PAD Trial is a Phase II multi-centered randomized clinical trial. Thirty-two participants with PAD will be randomized at one of two centers: Northwestern University (PI: MM McDermott, MD) and the University of Alabama (PI: Nicole Lohr MD, PhD) to either 660 nm light + home-based exercise or sham light + home-based exercise for four months. Both groups of participants will receive the same home-based high intensity walking exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

First, all participants will be age 50 and older. Second, all participants will have PAD. PAD will be defined as:

1. An ABI <= 0.90 at baseline.
2. Vascular lab evidence of PAD (such as a toe brachial pressure < 0.70 or an ankle brachial index less than or equal to 0.90), or angiographic evidence of PAD defined as at least 70% stenosis of an artery supplying the lower extremities.
3. An ABI of >0.90 and <= 1.00 who experience a 20% or greater drop in ABI in either leg after the heel-rise test.

Exclusion Criteria:

1. Above- or below-knee amputation
2. Critical limb ischemia defined as an ABI <0.30 or <0.40 with symptoms of rest pain
3. Wheelchair confinement or requiring a walker to ambulate
4. Walking is limited by a symptom other than PAD
5. Current foot ulcer on bottom of foot
6. Failure to successfully complete the study run-in
7. Planned major surgery, coronary or leg revascularization during the next four months
8. Major surgery, coronary or leg revascularization or major cardiovascular event in the previous three months
9. Major medical illness including lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent, unless the cancer is located in the lower extremities. Participants who require oxygen only at night may still qualify.]
10. Mini-Mental Status Examination (MMSE) score < 23
11. Non-English speaking
12. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
13. Visual impairment that limits walking ability.
14. Six-minute walk distance of <400 feet or >1700 feet.
15. Participation in a supervised treadmill exercise program or a cardiac rehabilitation program in previous three months or planning to begin a supervised treadmill exercise program or a cardiac rehabilitation program in the next five months.
16. Unwilling to avoid red light therapy outside of study participation.
17. Baseline blood pressure <100/45.
18. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Distance | Measured at baseline and 4-month follow-up
  Change in six-minute walk distance
Six-Minute Walk Distance | Measured immediately after the first light treatment (within 15 minutes after the first treatment, acute effect)
  Change in six-minute walk distance (acute effect)

SECONDARY OUTCOMES:
Six-Minute Walk Distance | Measured at 4-month follow-up, 24 hours after the final treatment
  Change in six-minute walk distance (chronic effect)
Gastrocnemius Perfusion | Measured at baseline and 4-month follow-up
  Changes in calf perfusion at 3 Tesla measured with arterial spin labeling with MRI and post-cuff occlusion hyperemia
Minutes of High Intensity Exercise | Measured at baseline and 4-month follow-up
  Change in minutes of high intensity exercise/week (measured by the ActiGraph activity monitor)
Mean Exercise Intensity | Measured at baseline and 4-month follow-up
  Change in mean exercise intensity (measured by the ActiGraph activity monitor)
Mean Exercise Intensity During Six-Minute Walk | Measured at baseline and 4-month follow-up
  Change in mean exercise intensity during the six-minute walk (measured by the ActiGraph activity monitor)
Walking Impairment Questionnaire Distance Score | Measured at baseline and 4-month follow-up
  Participant report of difficulty walking increasingly longer distances. Score range 0-100, 100 is best
PROMIS Mobility Score | Measured at baseline and 4-month follow-up
  PROMIS mobility score from administered PROMIS questionnaire. Score range is from zero to infinity and a higher score means a better outcome.

OTHER OUTCOMES:
Walking Impairment Questionnaire Speed Score | Measured at baseline and 4-month follow-up
  Participant report of ability to walking increasing number of stair flights (0-100 score, 100-best)
Walking Impairment Questionnaire Stair Climbing Score | Measured at baseline and 4-month follow-up
  Participant report of ability to walking increasing number of stair flights (0-100 score, 100-best)
Short-Form 36 (SF-36) Score (0-100 score, 100-best) | Measured at baseline and 4-month follow-up
  Change in score on the SF-36 from baseline to follow-up
Short Physical Performance Battery (SPPB) | Measured at baseline and 4-month follow-up
  SPPB range, range 0-12, 12-best
Plasma Nitrite | Measured before and within five minutes after the first light treatment at baseline
  Changes in plasma abundance of nitrite
Plasma Nitrite | Measured before and within five minutes after the final light treatment at 4-month follow-up
  Changes in plasma abundance of nitrite
Plasma Nitrosothiols | Measured before and within five minutes after the first light treatment at baseline
  Changes in plasma abundance of nitrosothiols
Plasma Nitrosothiols | Measured before and within five minutes after the final light treatment at 4-month follow-up
  Changes in plasma abundance of nitrosothiols
Gastrocnemius Muscle Capillary Density | Measured at baseline and 4-month follow-up
  Changes in gastrocnemius muscle capillary density
Gastrocnemius Muscle Myofiber Size | Measured at baseline and 4-month follow-up
  Changes in gastrocnemius muscle myofiber size
Gastrocnemius Muscle Citrate Synthase Activity | Measured at baseline and 4-month follow-up
  Changes in gastrocnemius muscle citrate synthase activity
Gastrocnemius Muscle Cytochrome C Oxidase Activity | Measured at baseline and 4-month follow-up
  Changes in gastrocnemius muscle cytochrome c oxidase activity
Gastrocnemius Muscle Abundance of Satellite Cells | Measured at baseline and 4-month follow-up
  Changes in gastrocnemius muscle abundance of satellite cells
Gastrocnemius Muscle Abundance of Myofibers with Central Nuclei | Measured at baseline and 4-month follow-up
  Changes in gastrocnemius muscle abundance of myofibers with central nuclei

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States